CLINICAL TRIAL: NCT01276587
Title: Pilot Study of Vitamin D Therapy to Prevent Respiratory Complications in Children With Sickle Cell Disease
Brief Title: Study of Vitamin D in Children With Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gary M Brittenham, MD (Other)
Responsible Party: Sponsor-Investigator, Gary M Brittenham, MD, James A. Wolff Professor of Pediatrics, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF2598
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2018-03

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; children; vitamin D; safety
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Oral vitamin D3 100,000 IU administered monthly for six months in children and adolescents with sickle cell disease
  Other Names: Vitamin D

SUMMARY:
This pilot study aims to answer the question whether monthly oral vitamin D3 supplementation, 100,000 IU, will be safe and effective in raising serum 25-hydroxyvitamin D (form of vitamin D measured in the blood) to levels considered sufficient (30 ng/mL) but well below the threshold for toxicity (150 ng/mL) in children with sickle cell disease. Information from this study will be crucial before we perform a larger clinical trial to determine the effects of vitamin D in reducing respiratory complications in patients with sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is a genetic red blood cell disorder that affects an estimated 89,000 Americans, predominantly those of African ancestry. The leading causes of morbidity and of death in sickle cell disease are respiratory complications, particularly a life-threatening lung disease unique to sickle cell disease called the "acute chest syndrome". An infectious trigger and a pro-inflammatory state appear to be critical mechanisms of the respiratory problems in sickling disorders. Emerging evidence that vitamin D has antimicrobial and anti-inflammatory functions in the respiratory tract, and the recognition of widespread vitamin D insufficiency in sickle cell children provide a compelling new rationale for vitamin D supplementation in sickle cell disease.

This will be an open label, single arm study to assess the efficacy and safety of oral vitamin D3 100,000 IU administered monthly for six months in children and adolescents with sickle cell disease. Twelve pediatric patients with sickle cell disease, 3-20 years old, will be recruited. The primary outcome measure (efficacy and safety) will be serum 25-hydroxyvitamin D concentration. Other safety measures will include serum calcium and urinary calcium and creatinine. Serial measurements of serum 25-hydroxyvitamin D, serum chemistries, and urinary calcium and creatinine will be performed at baseline entry, monthly for six months during treatment with vitamin D3, and at study exit. Other measures relevant to our planned Phase 2 clinical trial, including markers of bone turnover, immune function, and inflammation, will also be obtained at baseline, midpoint and exit. Recruitment and enrollment of subjects is expected to be for 3 months; study assessments will be for 7 months (1 month screening and 6 months treatment); and, the remaining 2 months will be devoted to data collation and analysis.

Study Procedures

Screening: After signing written informed consent by a parent or legal guardian (and assent, if applicable) or patient, eligible participants will undergo a screening examination including a standardized history and physical examination.

A venous blood sample will be obtained for baseline screening measures including serum 25-hydroxyvitamin D, serum chemistries, and urine calcium and creatinine. Within one month, eligible participants who do not have any of the exclusion criteria will return for enrollment in the pilot study.

Intervention: Participants will be seen monthly for administration of oral vitamin D3 100,000 IU under the direct observation by the Clinical Research Nurse. History and examination will be performed to capture symptoms and signs of adverse events. Questionnaires to collect data on vitamin D and calcium dietary intake and respiratory events will be administered. Venous blood and urine samples for study assessments (serum 25-hydroxyvitamin D, serum albumin, calcium and phosphate, urine calcium and creatinine) will be obtained at each visit prior to administration of study drug.

ELIGIBILITY:
Inclusion Criteria:

* patients with sickle cell disease
* 3 to 20 years old
* pregnant females with sickle cell disease are eligible

Exclusion Criteria:

* no informed consent or assent
* unable or unwilling to comply with requirements of the clinical trial
* participation in another clinical trial
* history of hypercalcemia or diagnosis of any medical condition associated with hypercalcemia, such as primary hyperparathyroidism, malignancy, familial hypocalciuric hypercalcemia, William's syndrome and other rare causes
* therapy with thiazide diuretics or lithium carbonate
* known renal or liver disease
* known malabsorption syndrome and inflammatory bowel disease
* chronic use of corticosteroids, excluding inhaled steroids
* current use of anticonvulsants (phenytoin, phenobarbital, carbamazepine)
* current intake of vitamin D and calcium supplements
* initiation of hydroxyurea or iron chelation therapy within the past 3 months
* serum 25hydroxyvitamin D >60 ng/mL

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret T Lee, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 3
  Unknown or Not Reported | 0
Serum 25-hydroxyvitamin D level [Mean (Standard Deviation); unit: ng/mL] | 10.5 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Serum 25-hydroxyvitamin D Concentration
Description: Serum 25-hydroxyvitamin D level was measured at 6 months.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Single Arm
Number analyzed (Participants) | 4
ng/mL
  Month 1 | 28.5 (6.19)
  Month 2 | 36.5 (7.94)
  Month 3 | 41.0 (9.38)
  Month 4 | 41.75 (8.88)
  Month 5 | 40.75 (11.93)
  Month 6 | 42.5 (9.95)

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes